CLINICAL TRIAL: NCT06599827
Title: Neoadjuvant Moderately Hypofractionated Radiotherapy Combined with Chemotherapy and Immunotherapy for High-risk PMMR/MSS Locally Advanced Rectal Cancer: a Prospective, Exploratory Phase II Trial（iMHRT-LARC）
Brief Title: Neoadjuvant Moderately Hypofractionated Radiotherapy Combined with Chemotherapy and Immunotherapy for High-risk LARC
Acronym: iMHRT-LARC
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Shanghai Zhongshan Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: B2024-271
Record Dates: First submitted 2024-09-05; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Rectal Cancer
Keywords: Moderately Hypofractionated Radiotherapy; Immunotherapy; Locally Advanced Rectal Adenocarcinoma; Chemotherapy
MeSH Terms: conditions — Rectal Neoplasms | interventions — Drug Therapy; Immunotherapy; Surgical Procedures, Operative

STUDY DESIGN:
Intervention Model Description: Patients will receive CapeOx chemotherapy, anti-PD-1 mAb immunotherapy, and moderately hypofractionated radiotherapy.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Experimental group (Experimental): This study examines combined radiotherapy, chemotherapy, and immunotherapy for high-risk locally advanced rectal cancer. After a week post-radiotherapy, patients start CapeOx chemotherapy with anti-PD-1 mAb. Surgery follows after 3 cycles of this regimen.
  Interventions: Radiation: moderately hypofractionated radiotherapy; Drug: chemotherapy; Drug: immunotherapy; Procedure: Total mesorectal excision (TME) surgery

INTERVENTIONS:
Radiation: moderately hypofractionated radiotherapy — 35 Gy in 10 fractions to mesorectal and metastatic lymph nodes, and 30 Gy in 10 fractions to pelvic lymphatic drainage area, weekly over 5 days at 3-3.5 Gy/day.
Drug: chemotherapy — CapeOx-Capecitabine 1000 mg/m² orally twice daily (days 1-14, every 21 days) + Oxaliplatin 130 mg/m² IV (day 1, every 21 days).
Drug: immunotherapy — Serplulimab 300 mg IV infusion on day 1 every 21 days.
Procedure: Total mesorectal excision (TME) surgery — Total mesorectal excision (TME) surgery assessment post 3 cycles of chemotherapy and immunotherapy; eligible patients undergo TME surgery.

SUMMARY:
This study aims to evaluate the effectiveness and safety of combining moderately hypofractionated radiotherapy with chemotherapy and anti-PD-1 antibodies as a neoadjuvant treatment for high-risk locally advanced rectal cancer.

DETAILED DESCRIPTION:
This study investigates a novel treatment approach involving moderately hypofractionated radiotherapy (3-3.5Gy×10) combined with chemotherapy and immunotherapy for patients with high-risk locally advanced rectal adenocarcinoma, aiming to optimize treatment efficacy and patient outcomes.

Neoadjuvant chemoradiotherapy followed by total mesorectal excision (TME) is the standard of care for locally advanced rectal cancer, improving surgical resection rates, local control, and sphincter preservation. Conventional long-course radiotherapy is the standard modality for neoadjuvant therapy, but it has drawbacks such as long treatment duration, high cost, and prolonged preoperative waiting time. Short-course radiotherapy, on the other hand, offers shorter treatment duration, lower cost, and shorter preoperative waiting time, but it is associated with higher rates of local recurrence. Immunotherapy has demonstrated promising anti-tumor activity in colorectal cancers with deficient mismatch repair (dMMR) and/or microsatellite instability-high (MSI-H) status, but its role in proficient mismatch repair (pMMR) and/or microsatellite stable (MSS) colorectal cancers remains unclear. However, studies have shown that the combination of chemoradiotherapy and immunotherapy can increase the pathologic complete response rate compared to chemoradiotherapy alone, suggesting that radiotherapy may serve as a stimulator of adaptive immunity and synergize with immunotherapy. Therefore, this study aims to explore the following regimen: neoadjuvant moderately hypofractionated radiotherapy at a dose of 3.5 Gy × 10 fractions to the tumors and 3 Gy × 10 fractions to the pelvic lymph node drainage area, combined with chemotherapy (capecitabine and oxaliplatin) and immunotherapy (Serplulimab).

This prospective, single-center, non-randomized Phase II trial is designed to explore the efficacy and safety of the treatment regimen. Patients will receive CapeOx chemotherapy, anti-PD-1 monoclonal antibody immunotherapy, and a course of moderately hypofractionated radiotherapy. The trial protocol prioritizes safety monitoring and efficacy assessments through standardized clinical and imaging evaluations.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 and ≤75 years.
2. MRI-confirmed rectal adenocarcinoma with the lower edge of the lesion ≤10cm from the anal verge.
3. Immunohistochemistry confirms proficiency in DNA mismatch repair (pMMR), or genetic testing confirms microsatellite instability-low (MSI-L) or microsatellite stable (MSS) status.
4. Pelvic MRI showing one of the following high-risk factors: cT4a/b; N2; extramural vascular invasion (EMVI+); mesorectal fascia involvement (MRF+); enlarged lateral lymph nodes.
5. ECOG performance status of 0-1.
6. No prior surgery, radiotherapy, chemotherapy, or targeted therapy.
7. Tolerable to radiotherapy, chemotherapy, and immunotherapy with laboratory results: WBC ≥4.0 × 10^9/L, platelets ≥100 × 10^9/L, hemoglobin ≥80g/L, ALT <2ULN, TB <35μmol/L, Scr <1.5ULN or creatinine clearance rate ≥50mL/min, TSH ≤ULN (if abnormal, consider T3 and T4 levels; if T3 and T4 are normal, patients can still be included).
8. Voluntary participation with signed informed consent.

Exclusion Criteria:

1. Distant metastases.
2. Stage I or II rectal cancer not requiring neoadjuvant therapy.
3. Severe cardiovascular, pulmonary, neurological, renal, gastrointestinal, or systemic diseases.
4. Untreated chronic hepatitis B carrier with HBV DNA >500 IU/ml, HCV RNA positive patients, except for inactive hepatitis B surface antigen carriers, stable hepatitis B (HBV DNA <500 IU/ml), and cured hepatitis C patients.
5. History of active autoimmune diseases or potential relapse of autoimmune diseases.
6. Patients who received corticosteroids (equivalent to prednisone >10mg/day) or other immunosuppressive therapy within 2 weeks prior to study drug administration.
7. History of thyroid dysfunction.
8. Severe chronic or active infections requiring systemic antifungal or antiviral therapy, including tuberculosis.
9. Known allergy or hypersensitivity to multiple drugs.
10. History of pelvic radiation.
11. History of inflammatory bowel disease.
12. Unwillingness to participate or sign informed consent.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Estimated)
Dates: Start 2024-09-20 (Estimated); Primary Completion 2026-09-20 (Estimated); Study Completion 2029-09-20 (Estimated)

PRIMARY OUTCOMES:
pathologic complete response (pCR) | 30-day
  Proportion of patients in whom no cancer cells are found in resected rectal tissue and regional lymph nodes upon pathological evaluation.

SECONDARY OUTCOMES:
disease-free survival (DFS) | 3-year
  DFS is defined as the time from randomization until disease recurrence or death from any cause.
event-free survival (EFS) | 3-year
  Time from treatment initiation to occurrence of any of the following: disease progression affecting surgery, post-operative disease progression or recurrence, or death from any cause.
objective response rate (ORR) | 3-month
  Proportion of patients showing partial or complete response to treatment, defined by RECIST v1.1 as ORR=(CR+PR)/ITT*100%.
overall survival (OS) | 3-year
  OS is defined as the time from randomisation to death.
adverse events | 3-year
  Incidence of adverse events: According to CTCAE 5.0.
Quality of Life (QoL)-LARS socre | 3-year
  LARS score questionnaire: A tool used to assess bowel function and quality of life after rectal surgery, focusing on symptoms like frequency of bowel movements, urgency, and incontinence. The score ranges from 0 to 42, with higher scores indicating more severe symptoms and a greater impact on quality of life.
Quality of Life (QoL)-Wexner score | 3-year
  Wexner score: Wexner score composed of five items (solid, liquid, gas, wears pad, and lifestyle alteration) and five frequencies, resulting in a total score ranging from 0 (perfect continence) to 20 (complete incontinence). The score includes pad usage and lifestyle alteration, providing a comprehensive assessment of the impact of fecal incontinence on a patient's daily life
Quality of Life (QoL)-FISI score | 3-year
  FISI score: The Fecal Incontinence Severity Index, a questionnaire that quantifies the impact of fecal incontinence on quality of life by assessing the frequency of incontinence episodes and related concerns. It includes four types of incontinence (gas, mucus, liquid, solid) and six frequencies, plus a "never" option. Each item is scored according to its frequency, and the total score ranges from 0 to 61, with higher scores indicating greater severity and impact on the patient's life.

CONTACTS AND LOCATIONS:
Overall Officials: Jian Wang, MD, Principal Investigator — Fudan University
Locations (1):
- Zhongshan Hospital, Fudan University, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No